CLINICAL TRIAL: NCT01445613
Title: CANOPY: Carotid Artery Stenting Outcomes in the Standard Risk Population for Carotid Endarterectomy
Brief Title: Carotid Artery Stenting Outcomes in the Standard Risk Population for Carotid Endarterectomy
Acronym: CANOPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-720
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Carotid Artery Disease; Stroke; Amaurosis Fugax; Transient Ischemic Attack (TIA)
Keywords: Carotid; Stent; Carotid Endarterectomy
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Amaurosis Fugax; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RX Acculink Carotid Stent System (RX Acculink) (Other): Those patients receiving the RX Acculink used with an Embolic Protection System (EPS) approved for use with RX Acculink.
  Interventions: Device: RX Acculink Carotid Stent System (RX Acculink)

INTERVENTIONS:
Device: RX Acculink Carotid Stent System (RX Acculink) — Those patients receiving the RX Acculink used with an Embolic Protection System (EPS) approved for use with RX Acculink.

SUMMARY:
The objective of the CANOPY trial is to assess the continued safety and effectiveness of the RX Acculink Carotid Stent System under commercial use in subjects at standard risk for adverse events from Carotid Endarterectomy (CEA) enrolled by physicians with a range of carotid stenting experience.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age.
2. Subject does not have any condition that limits their anticipated survival to less than 3 years.
3. Subject or a legally authorized representative must provide written informed consent prior to any trial related procedure.
4. Subjects with neurological symptoms within 180 days of the procedure and ≥ 70% stenosis of the common or internal carotid artery by ultrasound or ≥ 50% stenosis of the common or internal carotid artery by angiogram - OR-
5. Subjects without neurological symptoms within 180 days of the procedure and ≥ 70% stenosis of the common or internal carotid artery by ultrasound or ≥ 60% stenosis of the common or internal carotid artery by angiogram.
6. Subject with all the following target vessel characteristics:

   1. Discrete lesion in internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA).
   2. Vessel diameter ≥ 4.0 mm and ≤ 9.0 mm from reference or contralateral artery.
   3. Absence of excessive vessel tortuosity that would impede delivery of devices.
7. Subject must agree not to participate in any other clinical trial for a period of 1 year following the index procedure.

Exclusion Criteria:

1. Subjects with anatomic or clinical conditions which make them at high risk for adverse events from carotid endarterectomy (CEA).
2. Subject with Hgb <10.g/dl or platelet count < 125,000 µl or has heparin-associated thrombocytopenia. For subjects on Coumadin (Warfarin) and for subjects with a platelet or coagulation disorder: Has an international normalized ratio (INR) > 1.5.
3. Subject has active bleeding diathesis or coagulopathy or subject would refuse blood transfusions.
4. Subject is currently on a list for major organ transplantation (i.e., heart, lung, liver, kidney) or is being evaluated for such.
5. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
6. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1203 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Christopher Metzger, MD, Principal Investigator — Wellmont Holston Valley Medical Center
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for the CANOPY clinical trial started on October 11, 2011 and was completed on September 12, 2013. The enrollment goal (1200 subjects) was reached with a total of 1203 subjects enrolled at 97 clinical sites.
Pre-assignment Details: 3/1203 subjects who received a non-study stent, were excluded from the analysis. A total of 1200 subjects were included in the primary analysis population (Full analysis set (FAS)).
Period: 30-day Follow-up
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Started | 1200
Completed | 1165
Not Completed | 35
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 3
Not completed — Missed visit | 23
Not completed — Death | 3
Period: 1-year Follow-up
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Started | 1165
Completed | 1088
Not Completed | 77
Not completed — Withdrawal by Subject | 12
Not completed — Missed visit | 29
Not completed — Lost to Follow-up | 2
Not completed — Death | 30
Not completed — Physician Decision | 2
Not completed — Received a non-study stent | 2

BASELINE CHARACTERISTICS:
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.52 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 491
  Male | 709
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 10
  Asian | 14
  Black or African Heritage | 69
  Native Hawaiian or other Pacific Islander | 1
  White | 1083
  Hispanic or Latino | 30
  Refused to answer | 3
  Information not available | 3
Region of Enrollment [Number; unit: participants]
  United States | 1200

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Peri-procedural (Within 30 Days of the Procedure) Death and Stroke, Plus Ipsilateral Stroke Between Day 31 and 1 Year (365 Days)
Time Frame: 0 to 365 days
Population: FAS population
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
percentage of participants | 4.4 (0.60)

2. Secondary Outcome: Death and All Stroke
Time Frame: 30 Days
Population: FAS population. The number of participants analyzed includes subjects with data available at that time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1178
percentage of participants | 3.4 [2.44 to 4.60]

3. Primary Outcome: Freedom From Death and Stroke Within 30 Days and Ipsilateral Stroke Between 31 and 365 Days
Time Frame: 365 days
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
percentage of participants | 95.6

4. Secondary Outcome: Composite of Peri-procedural Death and Stroke by Symptomatic Status
Time Frame: 30 days
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Composite of Peri-procedural DS in the Symptomatic Group: Symptomatic subject: Subject with Amaurosis Fugax (a temporary (≤10 minutes) loss of vision in one eye due to insufficient blood flow to the retina), stroke or transient ischemic attack (TIA) (hemispheric or ocular) in the hemisphere supplied by the target vessel in the last 180-days prior to procedure.
- Composite of Peri-procedural DS in the Asymptomatic Group: Asymptomatic Subject: Subject does not have a history of symptoms, stroke or TIA (hemispheric or ocular/Amaurosis Fugax) in the hemisphere supplied by the target vessel in the last 180 days.
Arm/Group | Composite of Peri-procedural DS in the Symptomatic Group | Composite of Peri-procedural DS in the Asymptomatic Group
Number analyzed (Participants) | 335 | 865
percentage of participants | 5.8 [3.55 to 8.95] | 2.5 [1.53 to 3.74]

5. Secondary Outcome: Freedom From Death and Stroke Within 30 Days and Ipsilateral Stroke Through 1 Year by Symptomatic Status
Time Frame: 365 days
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- In Symptomatic Group: Symptomatic subject: Subject with Amaurosis Fugax (a temporary (≤10 minutes) loss of vision in one eye due to insufficient blood flow to the retina), stroke or TIA (hemispheric or ocular) in the hemisphere supplied by the target vessel in the last 180-days prior to procedure.
- In Asymptomatic Group: Asymptomatic Subject: Subject does not have a history of symptoms, stroke or TIA (hemispheric or ocular/Amaurosis Fugax) in the hemisphere supplied by the target vessel in the last 180 days.
Arm/Group | In Symptomatic Group | In Asymptomatic Group
Number analyzed (Participants) | 335 | 865
percentage of participants | 92.5 | 96.8

6. Secondary Outcome: Composite of Peri-procedural Death and Stroke by Age
Time Frame: 30 days
Population: FAS population. The number of participants analyzed includes subjects with data available at that time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- In Octogenarian Group: Octogenarian: A person with age >= 80 years.
- In Non-octogenarian Group: Non-octogenarian: A person who is less than 80 years old.
Arm/Group | In Octogenarian Group | In Non-octogenarian Group
Number analyzed (Participants) | 116 | 1062
percentage of participants | 3.4 [0.95 to 8.59] | 3.4 [2.39 to 4.66]

7. Secondary Outcome: Freedom From Death and Stroke Within 30 Days and Ipsilateral Stroke Through 1 Year by Age
Time Frame: 365 days
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | In Octogenarian Group | In Non-octogenarian Group
Number analyzed (Participants) | 118 | 1082
percentage of participants | 93.8 | 95.8

8. Secondary Outcome: Freedom From Clinically Driven Target Lesion Revascularization
Description: Target Lesion Revascularization (TLR) is designated as clinically driven if the subject has recurring symptoms or has become newly symptomatic and has stenosis >50% in the stented lesion, or is asymptomatic and has a stenosis of >80% in the stented lesion.
Time Frame: 30 days
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
percentage of participants | 99.9

9. Secondary Outcome: Freedom From Clinically Driven Target Lesion Revascularization
Description: as for outcome 8
Time Frame: 180 days
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
percentage of participants | 99.7

10. Secondary Outcome: Freedom From Clinically Driven Target Lesion Revascularization
Description: as for outcome 8
Time Frame: 365 days
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
percentage of participants | 99.3

11. Secondary Outcome: Clinical Success
Description: Clinical success is defined as the attainment of < 50% residual stenosis of the target lesion and absence of a death or stroke 30-day post-procedure.
Time Frame: 30 days
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Number analyzed (Participants) | 1200
percentage of participants | 96.4 [95.2 to 97.39]

ADVERSE EVENTS:
Time Frame: 365 Days
Arm/Group | RX Acculink Carotid Stent System (RX Acculink)
Serious Adverse Events (participants affected / at risk) | 266/1200
Other Adverse Events (participants affected / at risk) | 619/1200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RX Acculink Carotid Stent System (RX Acculink) (N=1200)
Hematoma (General disorders) | 1 — Access Site Complication
Infection At Insertion Site (General disorders) | 1 — Access Site Complication
Other: under access site complication (General disorders) | 1 — Access Site Complication
Allergic Reaction To Contrast (Immune system disorders) | 1
GI Bleed (Blood and lymphatic system disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 7 — Blood Dyscrasia
Bleeding (Blood and lymphatic system disorders) | 1 — Blood Dyscrasia
Coagulopathy (Blood and lymphatic system disorders) | 1 — Blood Dyscrasia
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Abnormal Lab Test (Cardiac disorders) | 1
Angina (Cardiac disorders) | 6
Arrhythmia (Includes Brady And Tachy) (Cardiac disorders) | 10
Coronary artery disease - Coronary stenosis (Cardiac disorders) | 5
Cardiac Arrest (Cardiac disorders) | 6
Congestive Heart Failure (Cardiac disorders) | 6
Dyspnea (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 7
Myocardial Infarction - Non Q wave (Cardiac disorders) | 3
Myocardial Infarction - Q wave (Cardiac disorders) | 2
Myocardial Infarction - Unknown (Cardiac disorders) | 3
Peripheral vascular disease (Cardiac disorders) | 1
Pain (Cardiac disorders) | 4
Surgery/Intervention Procedure (Cardiac disorders) | 4
Syncope (Cardiac disorders) | 2
Thrombosis (Cardiac disorders) | 1
Other (Cardiac disorders) | 1
Bleeding (Gastrointestinal disorders) | 3
Diverticulitis (Gastrointestinal disorders) | 1
GI Bleed (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Other (Gastrointestinal disorders) | 5
Hematuria (Renal and urinary disorders) | 2
Kidney Damage Due To Other (Renal and urinary disorders) | 2
Malignant (Renal and urinary disorders) | 1
Renal Artery Disease (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 3
Sepsis (Renal and urinary disorders) | 1
Surgery/Intervention Procedure (Renal and urinary disorders) | 1
Tumor (Renal and urinary disorders) | 1
Urinary Retension (Renal and urinary disorders) | 2
Urinary Tract Infection (Renal and urinary disorders) | 3
Other (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Wound Complication Or Wound Infection (Infections and infestations) | 1
Diabetes (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Sensory Deficit (Metabolism and nutrition disorders) | 1
Surgery/Intervention Procedure (Metabolism and nutrition disorders) | 1
Abnormal Lab Test (General disorders) | 1 — Miscellaneous
Anxiety (General disorders) | 1 — Miscellaneous
Claudication (General disorders) | 1 — Miscellaneous
Depression (General disorders) | 1 — Miscellaneous
Diarrhea (General disorders) | 1 — Miscellaneous
Other: under miscellaneous category (General disorders) | 7 — Miscellaneous
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Cellulitis (Musculoskeletal and connective tissue disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 2
Other (Musculoskeletal and connective tissue disorders) | 4
Bleeding (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 4
Delerium (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Mental Status Change (Nervous system disorders) | 3
Post Traumatic Hemorrage (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Speech Disturbance (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 5
Transient Ischemia Attack (Nervous system disorders) | 12
Vasovagal (Nervous system disorders) | 1
Visual Disturbances (Nervous system disorders) | 2
Other (Nervous system disorders) | 2
Anemia (General disorders) | 5 — Procedure Related
Arrhythmia (Includes Brady And Tachy) (General disorders) | 18 — Procedure Related
Bleeding (General disorders) | 2 — Procedure Related
Colitis (General disorders) | 1 — Procedure Related
Dissection (General disorders) | 3 — Procedure Related
Embolism (General disorders) | 1 — Procedure Related
Headache (General disorders) | 2 — Procedure Related
Hemiparesis (General disorders) | 1 — Procedure Related
Hypertension (General disorders) | 1 — Procedure Related
Hypotension (General disorders) | 60 — Procedure Related
Incisional Pain (General disorders) | 1 — Procedure Related
Infection At Insertion Site (General disorders) | 1 — Procedure Related
Ischemia (General disorders) | 1 — Procedure Related
No reflow (General disorders) | 1 — Procedure Related
Pain (General disorders) | 2 — Procedure Related
Pain At Insertion Site (General disorders) | 1 — Procedure Related
Pseudoaneurysm (General disorders) | 6 — Procedure Related
Pulmonary Edema (General disorders) | 1 — Procedure Related
Transient Ischemia Attack (General disorders) | 1 — Procedure Related
Vessel Trauma (General disorders) | 1 — Procedure Related
Viral, Bacterial And Fungal Infections (General disorders) | 2 — Procedure Related
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6
Other (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident - Major Hemorrhagic Ispilateral (Vascular disorders) | 3
Cerebrovascular accident - Major Hemorrhagic Non-Ispilateral (Vascular disorders) | 1
Cerebrovascular accident - Major Ischemic Ispilateral (Vascular disorders) | 8
Cerebrovascular accident - Major Ischemic Non-Ispilateral (Vascular disorders) | 2
Cerebrovascular accident - Minor Hemorrhagic Bilateral (Vascular disorders) | 1
Cerebrovascular accident - Minor Hemorrhagic Ispilateral (Vascular disorders) | 2
Cerebrovascular accident - Minor Hemorrhagic Non-Ispilateral (Vascular disorders) | 1
Cerebrovascular accident - Minor Ischemic Bilateral (Vascular disorders) | 3
Cerebrovascular accident - Minor Ischemic Ispilateral (Vascular disorders) | 23
Cerebrovascular accident - Minor Ischemic Non-Ispilateral (Vascular disorders) | 3
Aneurysm (Vascular disorders) | 1
Claudication (Vascular disorders) | 5
Deep vein thrombosis (Vascular disorders) | 1
Occlusion (Vascular disorders) | 3
Peripheral artery disease (Vascular disorders) | 3
Peripheral vascular disease (Vascular disorders) | 3
Restenosis (Vascular disorders) | 10
Thrombosis (Vascular disorders) | 1
Vascular (Vascular disorders) | 1
Other (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RX Acculink Carotid Stent System (RX Acculink) (N=1200)
Arrhythmia (Includes Brady And Tachy) (General disorders) | 107 — Procedure Related
Hypotension (General disorders) | 242 — Procedure Related
Bleeding (General disorders) | 4 — Access Site Complication
Ecchymosis/Bruising (General disorders) | 2 — Access Site Complication
Hematoma (General disorders) | 6 — Access Site Complication
Infection At Insertion Site (General disorders) | 1 — Access Site Complication
Pain (General disorders) | 2 — Access Site Complication
Pain At Insertion Site (General disorders) | 3 — Access Site Complication
Other (General disorders) | 2 — Access Site Complication
Allergic Reaction To Contrast (Immune system disorders) | 4 — Allergic Reaction
Rash (Immune system disorders) | 6 — Allergic Reaction
Other (Immune system disorders) | 5 — Allergic Reaction
Anemia (Blood and lymphatic system disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 3
Ecchymosis/Bruising (Blood and lymphatic system disorders) | 2
GI Bleed (Blood and lymphatic system disorders) | 2
Hematoma (Blood and lymphatic system disorders) | 7
Abnormal Lab Test (Blood and lymphatic system disorders) | 1 — Blood Dyscrasia
Anemia (Blood and lymphatic system disorders) | 13 — Blood Dyscrasia
Bleeding (Blood and lymphatic system disorders) | 2 — Blood Dyscrasia
Coagulopathy (Blood and lymphatic system disorders) | 1 — Blood Dyscrasia
Leukocytosis (Blood and lymphatic system disorders) | 1 — Blood Dyscrasia
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Abnormal Lab Test (Cardiac disorders) | 2
Angina (Cardiac disorders) | 13
Arrhythmia (Includes Brady And Tachy) (Cardiac disorders) | 42
Asystole (Cardiac disorders) | 3
Atrial Fibrillation (Cardiac disorders) | 1
CAD - Coronary stenosis (Cardiac disorders) | 5
Cardiac Arrest (Cardiac disorders) | 6
Congestive Heart Failure (Cardiac disorders) | 8
Dizziness (Cardiac disorders) | 1
Dyspnea (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 13
Hypotension (Cardiac disorders) | 23
Ischemia (Cardiac disorders) | 1
Myocardial Infarction - Non Q wave (Cardiac disorders) | 3
Myocardial Infarction - Q wave (Cardiac disorders) | 2
Myocardial Infarction - Unknown (Cardiac disorders) | 3
Peripheral vascular disease (PVD) (Cardiac disorders) | 1
Pain (Cardiac disorders) | 8
Spasm (Cardiac disorders) | 1
Surgery/Intervention Procedure (Cardiac disorders) | 5
Syncope (Cardiac disorders) | 2
Thrombosis (Cardiac disorders) | 1
Vasovagal (Cardiac disorders) | 1
Other (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Bleeding (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 1
Gastrointestinal (GI) bleed (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Other (Gastrointestinal disorders) | 6
Abnormal Lab Test (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Incontinence (Renal and urinary disorders) | 1
Kidney Damage Due To Other (Renal and urinary disorders) | 2
Malignant (Renal and urinary disorders) | 1
Renal Artery Disease (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 3
Sepsis (Renal and urinary disorders) | 1
Surgery/Intervention Procedure (Renal and urinary disorders) | 1
Tumor (Renal and urinary disorders) | 1
Urinary Retension (Renal and urinary disorders) | 5
Urinary Tract Infection (Renal and urinary disorders) | 6
Viral, Bacterial And Fungal Infections (Renal and urinary disorders) | 1
Other (Renal and urinary disorders) | 1
Cellulitis (Infections and infestations) | 2
Eye (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 3
Viral, Bacterial And Fungal Infections (Infections and infestations) | 3
Wound Complication Or Wound Infection (Infections and infestations) | 1
Abnormal Lab Test (Metabolism and nutrition disorders) | 1
Diabetes (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Joint pain (Metabolism and nutrition disorders) | 1
Sensory Deficit (Metabolism and nutrition disorders) | 1
Surgery/Intervention Procedure (Metabolism and nutrition disorders) | 1
Other (Metabolism and nutrition disorders) | 1
Abnormal Lab Test (General disorders) | 4
Anxiety (General disorders) | 1
Back Pain (General disorders) | 1
Bleeding (General disorders) | 1
Claudication (General disorders) | 2
Cough (General disorders) | 1
Depression (General disorders) | 1
Diarrhea (General disorders) | 1
Dizziness (General disorders) | 4
Edema (Non Pulmonary) (General disorders) | 1
Headache (General disorders) | 13
Hematoma (General disorders) | 1
Joint pain (General disorders) | 1
Nausea (General disorders) | 1
Pain (General disorders) | 14
Rash (General disorders) | 1
Vomiting (General disorders) | 2
Weakness (General disorders) | 3
Other (General disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Cellulitis (Musculoskeletal and connective tissue disorders) | 1
Headache (Musculoskeletal and connective tissue disorders) | 2
Hematoma (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain (Musculoskeletal and connective tissue disorders) | 6
Weakness (Musculoskeletal and connective tissue disorders) | 2
Other (Musculoskeletal and connective tissue disorders) | 5
Bleeding (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 7
Delerium (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 9
Mental Status Change (Nervous system disorders) | 6
Nausea (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 2
Numbness (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 2
Post Traumatic Hemorrage (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 5
Sensory Deficit (Nervous system disorders) | 1
Speech Disturbance (Nervous system disorders) | 7
Syncope (Nervous system disorders) | 10
Transient Ischemia Attack (Nervous system disorders) | 21
Vasovagal (Nervous system disorders) | 1
Visual Disturbances (Nervous system disorders) | 13
Weakness (Nervous system disorders) | 1
Other (Nervous system disorders) | 17
Abnormal Lab Test (General disorders) | 1 — Procedure Related
Access site event (General disorders) | 1 — Procedure Related
Allergic Reaction To Contrast (General disorders) | 1 — Procedure Related
Anemia (General disorders) | 15 — Procedure Related
Anxiety (General disorders) | 1 — Procedure Related
Asystole (General disorders) | 4 — Procedure Related
Back Pain (General disorders) | 3 — Procedure Related
Bleeding (General disorders) | 10 — Procedure Related
Colitis (General disorders) | 1 — Procedure Related
Dissection (General disorders) | 5 — Procedure Related
Ecchymosis/Bruising (General disorders) | 1 — Procedure Related
Embolism (General disorders) | 2 — Procedure Related
Eye (General disorders) | 1 — Procedure Related
Headache (General disorders) | 20 — Procedure Related
Hematoma (General disorders) | 19 — Procedure Related
Hemiparesis (General disorders) | 1 — Procedure Related
Hemorrhage (General disorders) | 1 — Procedure Related
Hypertension (General disorders) | 23 — Procedure Related
Incisional Pain (General disorders) | 1 — Procedure Related
Incontinence (General disorders) | 1 — Procedure Related
Infection At Insertion Site (General disorders) | 2 — Procedure Related
Ischemia (General disorders) | 1 — Procedure Related
Jaw Pain (General disorders) | 1 — Procedure Related
Mental Status Change (General disorders) | 2 — Procedure Related
Nausea (General disorders) | 18 — Procedure Related
Neuralgia (General disorders) | 1 — Procedure Related
No reflow (General disorders) | 1 — Procedure Related
Oozing (General disorders) | 1 — Procedure Related
Pain (General disorders) | 13 — Procedure Related
Pain At Insertion Site (General disorders) | 6 — Procedure Related
Paralysis (General disorders) | 1 — Procedure Related
Pseudoaneurysm (General disorders) | 8 — Procedure Related
Pulmonary Edema (General disorders) | 1 — Procedure Related
Renal Insufficiency (General disorders) | 1 — Procedure Related
Spasm (General disorders) | 4 — Procedure Related
Speech Disturbance (General disorders) | 1 — Procedure Related
Syncope (General disorders) | 1 — Procedure Related
Thrombosis (General disorders) | 2 — Procedure Related
Transient Ischemia Attack (General disorders) | 3 — Procedure Related
Urinary Retension (General disorders) | 2 — Procedure Related
Vasospasm (General disorders) | 4 — Procedure Related
Vasovagal (General disorders) | 3 — Procedure Related
Vessel Trauma (General disorders) | 1 — Procedure Related
Viral, Bacterial And Fungal Infections (General disorders) | 2 — Procedure Related
Visual Disturbances (General disorders) | 4 — Procedure Related
Vomiting (General disorders) | 3 — Procedure Related
Weakness (General disorders) | 2 — Procedure Related
Other (General disorders) | 11 — Procedure Related
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6
Viral, Bacterial And Fungal Infections (Respiratory, thoracic and mediastinal disorders) | 1
Other (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident (CVA) - Major Hemorrhagic Ispilateral (Vascular disorders) | 3 — Stroke
Cerebrovascular accident (CVA)-Major Hemorrhagic Non-Ispilateral (Vascular disorders) | 1 — Stroke
Cerebrovascular accident (CVA) - Major Ischemic Ispilateral (Vascular disorders) | 8 — Stroke
Cerebrovascular accident (CVA) - Major Ischemic Non-Ispilateral (Vascular disorders) | 2 — Stroke
Cerebrovascular accident (CVA) - Minor Hemorrhagic Bilateral (Vascular disorders) | 1 — Stroke
Cerebrovascular accident (CVA) - Minor Hemorrhagic Ispilateral (Vascular disorders) | 2 — Stroke
Cerebrovascular accident (CVA) - Minor Hemorrhagic Non-Ispilateral (Vascular disorders) | 1 — Stroke
Cerebrovascular accident (CVA) - Minor Ischemic Bilateral (Vascular disorders) | 3 — Stroke
Cerebrovascular accident (CVA) - Minor Ischemic Ispilateral (Vascular disorders) | 25 — Stroke
Cerebrovascular accident (CVA) - Minor Ischemic Non-Ispilateral (Vascular disorders) | 4 — Stroke
Aneurysm (Vascular disorders) | 3
Arrhythmia (Includes Brady And Tachy) (Vascular disorders) | 2
Claudication (Vascular disorders) | 6
Deep venous thrombosis (DVT) (Vascular disorders) | 2
Dissection (Vascular disorders) | 1
Occlusion (Vascular disorders) | 4
Peripheral artery disease (PAD) (Vascular disorders) | 3
Peripheral vascular disease (PVD) (Vascular disorders) | 4
Restenosis (Vascular disorders) | 10
Spasm (Vascular disorders) | 2
Surgery/Intervention Procedure (Vascular disorders) | 1
Syncope (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 2
Vascular (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 1
Vasovagal (Vascular disorders) | 1
Other (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days